CLINICAL TRIAL: NCT00192101
Title: Randomized Phase II Study of the Combination of Gemcitabine (Gemzar) Plus Cisplatin Single Dose Versus Split Dose in the Treatment of Patients With Locally Advanced or Metastatic Breast Cancer After Failure of Anthracyclines an/or Taxanes
Brief Title: Gemcitabine Plus Cisplatin Single Dose Versus Split Dose in the Treatment of Patients With Locally Advanced or Metastatic Breast Cancer After Failure of Anthracyclines and/or Taxanes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9590; B9E-SI-S371
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Cisplatin

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin

SUMMARY:
This is an open label, two arms, randomized, unblinded phase 2 study in patients with locally advanced or metastatic breast cancer who have been previously treated with anthracycline with/without taxane based regimen in the adjuvant/neoadjuvant or 1st line metastatic setting. Gemcitabine will be administered via intravenous infusion over approximately 30 minutes at a dose of 1250mg/m2 on days 1 and 8 of each 21-day cycle. In arm A:Cisplatin will be given via intravenous infusion over approximately 60-120 minutes at a dose of 70 mg/m2 on Day 1 of each 21-day cycle. The investigator may attempt to give Cisplatin with at least one liter of fluids for hydration and on an outpatient basis.

Patients will remain in the study until disease progression or when a maximum of six cycles have been administered. Study therapy may continue until:

* There is evidence of progressive disease
* The patient experiences unacceptable toxicity.
* The investigator decides that the patient should be discontinued.
* The patient requests discontinuation
* The patient has received 6 cycles of the regimen (if the physician decides to continue after 6 cycles-this will be done after consultation with the sponsor)
* Discontinuation from study therapy is indicated according to the additional guidelines described in the protocol After patients discontinue from study therapy, they proceed to the post-study follow up phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of breast carcinoma with evidence of unresectable, locally recurrent, or metastatic disease. Lesions should not be amenable to surgery or radiation of curative intent.
* Presence of metastatic or local-regional recurrent disease, according to the American Joint Committee on Cancer
* Uni-dimensionally measurable lesions with clearly defined margin that are clearly measurable by following methods according to computerized tomography (CT), Chest x-ray or clinical examination, according to RECIST criteria
* Patients with unresectable, locally recurrent or metastatic breast cancer who, were pre-treated with anthracyclines with/without taxanes (paclitaxel, docetaxel)containing chemotherapy either in neoadjuvant/adjuvant or 1st line metastatic setting will be enrolled into the study. Prior chemotherapy has to be terminated 4 weeks prior. Study randomization and disease progression under this therapy has to be documented, also patients must have completely recovered from all acute chemotherapy related toxicities (with exception of alopecia).

Prior radiotherapy must be completed at least 30 days before study entry. Patients must have recovered from the acute toxic effects of the treatment prior to study enrollment (except for alopecia). Lesions that have been radiated cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.

Exclusion Criteria:

* Have received treatment within the last 30 days with an investigational drug for any indication before study entry.
* Concurrent administration of other tumor therapy, including cytotoxic chemotherapy, surgery of cancer, radiotherapy, hormonal therapy and immunotherapy (including Herceptin)
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy, unless adequately treated.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment(except in situ carcinoma of cervix or adequately treated basal cell carcinoma of skin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-10; Study Completion 2005-07

PRIMARY OUTCOMES:
Overall response rates of the combination of gemcitabine and cisplatin in patients with locally advanced or metastatic breast cancer who have been previously treated with anthracycline with/without taxane based regimen
in the adjuvant/neoadjuvant or 1st line metastatic setting for each treatment arm separately.

SECONDARY OUTCOMES:
To characterize the quantitative and qualitative toxicity of gemcitabine-cisplatin patient population for each treatment arm separately;Relative dose intensity of gemcitabine and cisplatin for each treatment arm separately
Rate of dose modifications (omissions, reductions, delays) for each treatment arm separately;Time to progression for each treatment arm separately;Duration of response for each treatment arm separately;1-year survival in each treatment arm separately
Overall survival in each treatment arm separately;To assess the medical resources utilization with the combination in each treatment arm separately

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Jeddah, Saudi Arabia